CLINICAL TRIAL: NCT00004994
Title: A Study Comparing Quality of Life in Patients Undergoing a Non-Myeloablative Versus a Myeloablative Peripheral Blood Stem Cell Transplant for Hematological Diseases
Brief Title: Comparison of Quality of Life in Patients Undergoing More Intensive Versus Less Intensive Chemotherapy and Radiation Preceding a Bone Marrow Transplant
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 000002; 00-CC-0002
Record Dates: First submitted 2000-03-22; First posted 2000-03-23 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2004-10

CONDITIONS: Bone Marrow Transplantation
Keywords: Allogeneic Transplant; Function; Mini-Transplant; Physical Symptoms; Symptom Distress

SUMMARY:
This study will examine the quality of life of patients undergoing bone marrow transplantation to treat a blood disease. It will look at how this therapy affects many areas of life, including for example, personal relationships, work, and general emotional state. The information gained may lead to improved ways of dealing with problems that may arise before or during treatment.

Patients receiving bone marrow stem cells donated by a family member may participate in this study. They will be interviewed before treatment begins and will complete questionnaires at the following intervals:

1. day of admission to the hospital
2. day of the transplant
3. 30 days after the transplant
4. 100 days after the transplant
5. 1 year after therapy
6. 2 years after therapy

All questionnaires to be completed after discharge from the hospital will be scheduled during a regular follow-up visit. Each questionnaire takes about 15 to 20 minutes to complete. The information provided is confidential and will not be shared.

DETAILED DESCRIPTION:
Clinical research in blood stem cell and bone marrow transplantation documents improvements in disease free intervals, disease free survival, and the severity of treatment related toxicities. However, it is important for patients and families to know the quality of life (QOL) they can expect following an allogeneic transplant. In this longitudinal study we will compare the QOL of patients undergoing a non-myeloablative allogeneic peripheral blood stem cell transplant (A-PBSCT) prospectively with that of a myeloablative A-PBSCT. Subjects (n=106) over the age of 18 will be enrolled. Measures of quality of life (Medical Outcomes Study Short Form-MOS SF-36 and Functional Assessment of Cancer Therapy-General and Bone Marrow Transplant - FACT-G and FACT-G/BMT) and symptom distress (Symptom Distress Scale - SDS) will be administered prior to transplant (baseline) and at set interval post transplant. Data will be analyzed using repeated measures analysis of variance and regression analysis.

ELIGIBILITY:
INCLUSION CRITERIA:

Male or female subjects 18 years of age or older.

Able to read English or Spanish.

Hematological disease requiring A-PBSCT.

Signed informed consent for QOL study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 106
Dates: Start 1999-10; Study Completion 2004-10

CONTACTS AND LOCATIONS:
Locations (1):
- Warren G. Magnuson Clinical Center (CC), Bethesda, Maryland, United States

REFERENCES:
- [Background] Andrykowski MA, Henslee PJ, Farrall MG. Physical and psychosocial functioning of adult survivors of allogeneic bone marrow transplantation. Bone Marrow Transplant. 1989 Jan;4(1):75-81. PMID 2647190
- [Background] Andrykowski MA, Altmaier EM, Barnett RL, Otis ML, Gingrich R, Henslee-Downey PJ. The quality of life in adult survivors of allogeneic bone marrow transplantation. Correlates and comparison with matched renal transplant recipients. Transplantation. 1990 Sep;50(3):399-406. doi: 10.1097/00007890-199009000-00009. PMID 2402788
- [Background] Baker F, Wingard JR, Curbow B, Zabora J, Jodrey D, Fogarty L, Legro M. Quality of life of bone marrow transplant long-term survivors. Bone Marrow Transplant. 1994 May;13(5):589-96. PMID 8054912